CLINICAL TRIAL: NCT03288753
Title: Comparison of Patient Satisfaction and Audiological Performance Between Neuro 1 and Neuro 2 Speech Processors
Brief Title: Comparison Between Neuro 1 and Neuro 2 Cochlear Implant Speech Processors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIC_14
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Sensorineural Hearing Loss; Cochlear Hearing Loss
Keywords: Cochlear implant
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Noise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adults and children above 14 years old (Experimental): Visit 1:
  Satisfaction questionnaire on Neuro 1 Speech intelligibility in quiet on Neuro 1 Speech intelligibility in noise on Neuro 1 VRB (Vocale Rapide dans le Bruit) on Neuro 1
  Visit 2 (15 days after V1):
  Satisfaction questionnaire on Neuro 2 Speech audiometry in quiet on Neuro 2 Speech audiometry in noise on Neuro 2 VRB (Vocale Rapide dans le Bruit) on Neuro 2
  Visit 3 (3 months after V2):
  Satisfaction questionnaire on Neuro 2 Speech audiometry in quiet on Neuro 2 Speech audiometry in noise on Neuro 2 VRB (Vocale Rapide dans le Bruit) on Neuro 2
  Interventions: Other: Satisfaction questionnaire; Behavioral: Speech intelligibility in quiet; Behavioral: Speech intelligibility in noise; Behavioral: VRB (Vocale Rapide dans le Bruit)
- children up to 14 years old (Experimental): Visit 1 Satisfaction questionnaire on Neuro 1
  Visit 2 (15 days after V1):
  Satisfaction questionnaire on Neuro 2
  Visit 3 (3 months after V2):
  Satisfaction questionnaire on Neuro 2
  The questionnaires have to be filled in by the parents. The child can participate in the completion of the questionnaire if he is willing and understands the questions.
  Interventions: Other: Satisfaction questionnaire

INTERVENTIONS:
Other: Satisfaction questionnaire — Participants have to complete a satisfaction questionnaire on the Neuro 1 or 2 processor.
Behavioral: Speech intelligibility in quiet — The speech material corresponds to the lists of Lafon designed for cochlear implant patients. Each lists contains 17 monosyllabic words. Speech comprehension is evaluated by the percentage of correct words and the percentage of correct phonemes. Speech signals are presented at 65 dB SPL. 2 lists of 17 words are presented. At visit 1, the participants wear the sound processor Neuro 1. At visits 2 and 3, the participants wear the Neuro 2.
  Arms: Adults and children above 14 years old
Behavioral: Speech intelligibility in noise — The speech material corresponds to the lists of Lafon designed for cochlear implant patients. Each lists contains 17 monosyllabic words. Speech comprehension is evaluated by the percentage of correct words and the percentage of correct phonemes. Speech signals are presented at 65 dB SPL. 2 lists of 17 words are presented. The noise corresponds to a cocktail party presented at +10 dB SNR (Speech on Noise Ratio). At visit 1, the participants wear the sound processor Neuro 1. At visits 2 and 3, the participants wear the Neuro 2.
  Arms: Adults and children above 14 years old
Behavioral: VRB (Vocale Rapide dans le Bruit) — Speech intelligibility in noise measured with the test VRB (Vocale Rapide dans le Bruit, French version of the Quick Sin). This test measures the SNR (Signal to Noise Ratio) at which the listeners understand half of the words of a sentence correctly. The outcome measure is in dB. 3 lists are presented. Speech signals are presented at 60 dB SPL.
  Other Names: french Quick SIN
  Arms: Adults and children above 14 years old

SUMMARY:
The present study aims to evaluate patient satisfaction and audiological performance with their current cochlear implant speech processor, the Neuro 1, and to compare it with the satisfaction and performance obtained with the new speech processor, the Neuro 2.

DETAILED DESCRIPTION:
Nowadays, cochlear implants (CI) are successfully used to rehabilitate severe to profound sensorineural hearing loss. Oticon Medical recently developed a new cochlear implant system, including a new implantable internal part (Neuro Zti) and a new speech processor (Neuro 1). This new speech processor automatically detects and adapts to the sound environment, increasing the ease of listening in all situations. A second version of this speech processor has very recently been developed, called the Neuro 2. The Neuro 1 and 2 share the same signal processing characteristics and the "sound" delivered to the patient is similar. However, the Neuro 2 offers better ergonomics (smaller size and weight, rechargeable batteries…). Some improvements available on the Neuro 2 may be particularly interesting for children.

The aim of the present study is twofold: 1. Compare the satisfaction of adult and pediatric users for the speech processor Neuro 1 with their satisfaction for the Neuro 2, and 2. Show that audiological outcomes are at least as good for the Neuro 2 than for the Neuro 1.

The participants come at the hospital for three visits. The Neuro 1 is evaluated during the first visit (V1). Evaluation of the Neuro 2 takes place during the second (V2, 15 days after V1) and the third (V3, 3 months after V2).

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* Native French speaker or fluent French speaker
* Patient already fitted with one or two speech processor Neuro 1 for at least 5 months

Exclusion Criteria:

* vulnerable patients, at the exception of children (pregnant women, persons under guardianship)
* No Social security affiliation
* non-compliant patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
Satisfaction questionnaire | 15 minutes
  The listener has to rate his appreciation of the Neuro 1 and Neuro 2 device and the sound quality on 7 points scale. The outcome measure corresponds to averaged score. The questionnaire has been developed by Oticon Medical to investigate satisfaction patient for their current and future speech processors. This questionnaire is not validated in the literature.

SECONDARY OUTCOMES:
Speech comprehension in quiet | 15 mins
  The speech material corresponds to the lists of Lafon designed for cochlear implant patients. Each lists contains 17 monosyllabic words. Speech comprehension is evaluated by the percentage of words and the percentage of phonemes correctly repeated. This double scoring is used to avoid floor or ceiling effects that could happen with only one of these measures.
Speech comprehension in Noise | 15 mins
  The speech material corresponds to the lists of Lafon designed for cochlear implant patients. Each lists contains 17 monosyllabic words. Speech comprehension is evaluated by the percentage of words and the percentage of phonemes correctly repeated. This double scoring is used to avoid floor or ceiling effects that could happen with only one of these measures.
French Quick Sin | 5 mins
  This test measures the SNR (Signal to Noise Ratio) at which the listeners understand half of the words of a sentence correctly. The outcome measure is in dB.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Vincent, MD, PROF, Principal Investigator — Hôpital Roger Salengro CHRU de Lille
Locations (9):
- France (9):
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Roger Salengro, Lille
  - Hôpital Edouard Herriot, Lyon
  - CHRU de Nancy Hôpital central, Nancy
  - CHU de Nantes Hôtel-Dieu, Nantes
  - CHU Nice - Institut Universitaire de la Face et du Cou, Nice
  - Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice
  - Hôpital Pitié Salpêtrière - APHP, Paris
  - Hôpital Necker-Enfants Malades, Paris

IPD SHARING:
Plan to Share IPD: No